CLINICAL TRIAL: NCT06575023
Title: Tamponade vs Partial Myometrial Resection of Lower Uterine Segment in Management of Placenta Accreta Spectrum Cases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Nabil Abdelrahman, DR, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: management of placenta accreta
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tamponade of lower uterine segmentin managment of placenta accreta spectrum cases (Active Comparator): usage of tamponade of the lower uterine segment in managment of placnta accreta spectrum cases
  Interventions: Procedure: Tamponade of lower uterine segment in management of placenta accreta spectrum cases
- partial myometrial resection of lower uterine segment in management of placenta accreta spectrum (Active Comparator): partial resection of lower uterine segment myometrium
  Interventions: Procedure: partial myometrial resection of lower uterine segment in management of placenta accreta spectrum cases

INTERVENTIONS:
Procedure: Tamponade of lower uterine segment in management of placenta accreta spectrum cases — To compare the efficacy of lower uterine tamponade and partial lower myometrial resection in the management of intraoperative bleeding in cases with placenta accreta spectrum
  Arms: tamponade of lower uterine segmentin managment of placenta accreta spectrum cases
Procedure: partial myometrial resection of lower uterine segment in management of placenta accreta spectrum cases — tamponade vs partial myomertial resection of lower uterine segment in managment of placenta accreta spectrum cases
  Arms: partial myometrial resection of lower uterine segment in management of placenta accreta spectrum

SUMMARY:
To compare the efficacy of lower uterine tamponade and partial lower myometrial resection in the management of intraoperative bleeding in cases with placenta accreta spectrum .

DETAILED DESCRIPTION:
Placenta accreta spectrum (PAS) represents the spectrum of clinical conditions when part or whole of the placenta becomes abnormally adherent or invades the myometrium (1-2). Over the last 40 years, caesarean delivery rates around the world have risen from less than 10% to over 30%, and almost simultaneously a 10-fold increase in the incidence of PAS (3). PAS is one of the most dangerous conditions of the pregnancy as it is significantly associated with maternal morbidity and mortality (4).

Ultrasound imaging is the most commonly used technique to diagnose PAS disorders prenatally. There is also wide variation globally on the management of PAS disorders, with some centres opting for a radical approach, whereas others have proposed a range of conservative approaches (5).

The conservative approaches include one-step conservative surgery, leaving the placenta in situ, the Triple-P procedure, and transverse B-Lynch suture (1). Several techniques have been described for controlling massive bleeding associated with placenta previa caesarean sections ,including uterine packing with gauze ,balloon tamponades ,the B-Lynch suture,insertion of parallel vertical compression sutures, a square suturing technique and embolization or ligation of the uterine and internal iliac arteries , but there is awide variation in the success rate of these maneuvers. Over-sewing of the bleeding site is the most common procedure used for PPH management, but in many cases, the bleeding points located in the lower segment and cervical canal are too deep and their locations are unclear because of the severity of the bleeding(

ELIGIBILITY:
Inclusion Criteria:

* 1-Pregnant women with placenta previa /PAS diagnosed before delivery (by ultrasound and Doppler examination) .

  2 - Gestational age starting from 28 weeks onwards. 3- Women with at least 1 previous hysterotomy (e.g. Caesarean deliveries, myomectomy) 4- Elective or emergent Caesarean deliveries

Exclusion Criteria:

* A pre-existing decision of performing intrapartum hysterectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
amount of intraopertive blood loss. | 2 years
  compare of amount of blood loss between two methods by adding collected blood in suction apparatus in milliliters to amount of biood in the soaked towels

SECONDARY OUTCOMES:
ICU admission | 2 years
  yes or no admission number of days if there is ICU admission cause of admission
Re exploration | 2 years
  if there is exploration or no cause of re-exploration outcome of re-exploration
drop of HB level postoperative | 2 years
  result of substitution of HB level postoperative from preoperative in gmldl
blood transfusion | 2 years
  amount of transfused blood units

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sentilhes L, Goffinet F, Kayem G. Management of placenta accreta. Acta Obstet Gynecol Scand. 2013 Oct;92(10):1125-34. doi: 10.1111/aogs.12222. PMID 23869630